CLINICAL TRIAL: NCT02590211
Title: Poker, Skills and Associated Problems (PERHAPS). Controlled Experimental Single Centre Study of Poker Players: Study of the Cognitive Mechanisms Underlying Poker Skills and of the Specificity of Poker-related Problems
Brief Title: Poker, Skills and Associated Problems
Acronym: PERHAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC14_0036
Record Dates: First submitted 2015-10-06; First posted 2015-10-28 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Pathological Gambling
Keywords: experimental study; cognitive mechanisms; poker; cognitive remediation therapy
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- non-poker players (Other): (control group)
  Interventions: Behavioral: cognitive, emotional and clinical assessment
- expert unproblematic poker players (Other): (comparator)
  Interventions: Behavioral: cognitive, emotional and clinical assessment
- pathological poker players (Other): (comparator)
  Interventions: Behavioral: cognitive, emotional and clinical assessment

INTERVENTIONS:
Behavioral: cognitive, emotional and clinical assessment — Cognitive and emotional assessment: Posner paradigm applied to emotional information (attention and emotional perception abilities), the modified Wisconsin Card Sorting Test (mental flexibility), the Hayling Sentence Completion Task (verbal inhibition), the Go - No Go test (motor inhibition) and the expressive suppression method (facial expression inhibition) Clinical assessment: gambling course and habits, level of cognitive distortions, control attribution (locus of control), social phobia, motivation for gambling, impulsivity, co-addictions, coping and gambling related-damage

SUMMARY:
The PERHAPS project aims to fill two gaps in the scientific literature: on the one hand, studying the clinical and cognitive particularities of poker-related problems, and on the other hand, studying poker skill as a combination of multiple cognitive and emotional abilities. The underlying clinical aim is to develop a cognitive remediation therapy program dedicated to pathological gamblers.

DETAILED DESCRIPTION:
In the literature, although compulsive poker players undoubtedly share similarities with the compulsive gamblers of other gambling games, clinicians have observed significant specificities in these patients, in terms of personality profile, gaming practices and associated troubles. These specificities could influence the effectiveness of treatment and prevention strategies in many ways. However, there are very few studies focused on the specific poker-related problems, particularly compared to other practices.

Furthermore, skill at poker has often been treated as a unique and general ability. This binary vision is now considered widely insufficient and most researchers recommend exploring the individual cognitive abilities at play in poker skill. To the investigators knowledge, no study has done this to date.

Consequently, the PERHAPS project aims to fill two gaps in the scientific literature: on the one hand, studying the clinical and cognitive particularities of poker-related problems, and on the other hand, studying poker skill as a combination of multiple cognitive and emotional abilities.

Three profiles of poker players will be studied, depending on their gambling practices and whether or not they are addicted: a control group of 30 non-poker players, a group of 30 expert unproblematic poker players, and a group of 30 pathological poker players.

The three groups will be compared with one another on:

* Cognitive and emotional abilities (for expert players) or deficits (for pathological gamblers)
* Clinical particularities of poker-related problems

Secondarily (ancillary study), pathological poker gamblers will be compared with pathological gamblers of other gambling games (pure chance games n=30 and quasi-skill games n=30).

The PERHAPS project aims to improve knowledge of gambling addiction, particularly as regards poker, in order to optimise prevention and care strategies. The clinical aim is especially to construct a cognitive remediation therapy program. It also intends to discuss the legal framework applied to poker under the gambling regulation.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years
* good understanding of French, literate
* correct level of vision and hearing
* specific inclusion criteria for each group include frequency and length of poker practice, DSM-5 doagnostic criteria for gambling disorder

Exclusion Criteria:

* protected adults
* important cognitive deficit (assessed by the MMSE)
* psychotic syndrome whole life
* other psychiatric disorders (mood disorders, anxiety disorders) and addictive disorders (disorders related to the use of alcoholic or other substances, excluding nicotine) that are present and not stabilized
* unstable endocrine disorders
* significant neurological disorders (such as head injuries (except mild), neurodegenerative diseases, unbalanced epilepsy, mental retardation, etc.)
* psychoactive use (before participation)
* color blindness
* cardiac disorders
* electronic implants

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
attention and emotional perception performances | only one assessment so at baseline
  Modified Posner paradigm Performances will be compared between pathological poker players and non-poker players (to identify cognitive deficits in pathological players compared to baseline level) and between pathological poker players and expert unproblematic poker players (to identify cognitive deficits in pathological players compared to a gambler level)
mental flexibility performances | only one assessment so at baseline
  Wisconsin Test (M-WCST) Performances will be compared between pathological poker players and non-poker players (to identify cognitive deficits in pathological players compared to baseline level) and between pathological poker players and expert unproblematic poker players (to identify cognitive deficits in pathological players compared to a gambler level)
inhibition performances | only one assessment so at baseline
  Evaluation of inhibition at verbal level: Hayling sentence Completion Task Performances will be compared between pathological poker players and non-poker players (to identify cognitive deficits in pathological players compared to baseline level)
inhibition performances | only one assessment so at baseline
  Evaluation of inhibition at motor level : Go-No Go Task Performances will be compared between pathological poker players and non-poker players (to identify cognitive deficits in pathological players compared to baseline level)
inhibition performances | only one assessment so at baseline
  Evaluation of inhibition et expressive level : suppressive expression method Performances will be compared between pathological poker players and non-poker players (to identify cognitive deficits in pathological players compared to baseline level)

SECONDARY OUTCOMES:
gambling course and habits | only one assessment so at baseline
  Standardized maintenance grid. The interview allows you to explore gambling habits, possible abstinence periods, different games the game of choice, current practice, damage and the quality of shoring, and resources.
control attribution (locus of control) | only one assessment so at baseline
  three-dimensional control location scale of Levenson (IPAH)
level of cognitive distortions, | only one assessment so at baseline
  clinical questionnaires : Gambling Related Cognitions Scale (GRCS)
level of social phobia | only one assessment so at baseline
  clinical questionnaires : social phobia questionnaire Leibowitz,
motivation for gambling | only one assessment so at baseline
  clinical questionnaires : Gambling motivation questionnaire Reasons Questionnaire (GMQ)
impulsivity profile | only one assessment so at baseline
  clinical questionnaires : Impulsive Behavior Scale
psychiatric and addictive comorbidities | only one assessment so at baseline
  clinical questionnaires : Mini International Neuropsychiatric Interview (MINI)
coping and gambling related-damage | only one assessment so at baseline
  clinical questionnaires : COPE Brief Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: inclusion advertising — http://www.ifac-addictions.fr/participer-a-une-etude-3.html